CLINICAL TRIAL: NCT02350647
Title: TWO-ARM, SINGLE BLIND, RANDOMIZED POST-MARKET STUDY ON THE USE OF HEALICOIL™ REGENESORB SUTURE ANCHOR IN THE REPAIR OF TEARS OF THE ROTATOR CUFF
Brief Title: Suture Anchor Comparison in Rotator Cuff Repairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00031426
Record Dates: First submitted 2014-09-10; First posted 2015-01-30 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Rotator Cuff Injury
Keywords: Rotator cuff; Ossification; Suture anchors
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEALICOIL Regenesorb (Experimental): Suture anchor for rotator cuff repair
  Interventions: Device: Suture Anchor HEALOCOIL
- Twinfix Ultra HA (Active Comparator): Suture anchor for rotator cuff repair
  Interventions: Device: Suture anchor Twinfix Ultra HA

INTERVENTIONS:
Device: Suture Anchor HEALOCOIL — Rotator cuff tears will be repaired intraoperatively using suture anchors
  Arms: HEALICOIL Regenesorb
Device: Suture anchor Twinfix Ultra HA
  Arms: Twinfix Ultra HA

SUMMARY:
Patients will be randomized to receive HEALICOIL™ REGENESORB (the study anchor) or TWINFIX Ultra HA, a similar comparative product, for use in the repair of their shoulder injury. They will be asked to complete questionnaires throughout the study and will receive an MRI, CT and multiple ultrasound images. The MRIs and radiographs will be used to assess bony ingrowth at the repair site, and the ultrasound to assess repair success rate of the rotator cuff. The clinical and radiological outcomes will be compared between the study and control groups. It is hypothesized that there will be 85% high quality ossification at anchor site for HEALICOIL REGENESORB and 49.9% high quality ossification for TWINFIX Ultra HA at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 35 to 75 years at the time of surgery.
* Willing and able to give voluntary informed consent to participate in this investigation.
* Full thickness tear of the rotator cuff
* Tear requires repair within one year of initial diagnosis.
* Tear must be anatomically repairable (must be able to get tendon back to the medial position on the footprint and at least back to the tuberosity).
* Willing and able, in the opinion of the Investigator, to cooperate with study procedures, and willing to return to study site for all required post-operative study visits.

Exclusion Criteria:

* Evidence of acute trauma including fracture or dislocation of the shoulder joint.
* Chronic retraction.
* Evidence of active infection, osteomyelitis, sepsis or distant infection, which could spread to the index joint.
* Subject has had previous rotator cuff, arthroplasty or fracture procedures on the operative shoulder.
* Subject has had acromioplasty or diagnostic arthroscopy on the operative shoulder within one (1) year prior to scheduled surgery date.
* Evidence of osteomalacia or other metabolic bone disorder(s), which may impair bone or soft tissue function.
* Evidence of other significant shoulder pathology including (Type II-IV lesion, Bankart lesion, Hill Sachs lesion).
* Patient has grade 4 changes to articular cartilage in operative shoulder
* Inflammatory arthropathies.
* Significant muscle paralysis of the shoulder girdle.
* Painful pathologies of the cervical spine.
* Comminuted bone surface, which would compromise secure anchor fixation.
* Non-surgical rotator cuff associated treatment, such as corticosteroid injection, within one (1) month prior to scheduled surgery date.
* Participating in another investigational trial or ongoing study that would interfere with the assessment of the primary and secondary outcomes.
* Female patient who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods.
* Major psychiatric illness, developmental handicap or inability to read and understand the English language.
* Major medical illness that would preclude undergoing surgery.
* Known to be involved in any active injury litigation claims relating to the study shoulder.
* Unwilling or unable to be assessed according to study protocol for two years following surgery.
* Patient requires a concomitant SLAP repair procedure in operative shoulder.
* Surgeon plans to use a Platelet Rich Plasma product or another therapy intended to augment healing of the rotator cuff in the study procedure.
* Protocol specified surgical technique cannot be followed for this subject.
* Rotator cuff repair will be done via open (as opposed to arthroscopic) procedure.
* Any other reason (in the judgment of the investigator).

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Tolan, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Twinfix Ultra HA: Suture anchor for rotator cuff repair
  Suture anchor Twinfix Ultra HA
Period: Overall Study
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
Started | 32 | 32
Completed | 26 | 26
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Full Range); unit: years] | 60 [41 to 73] | 57 [41 to 72] | 59 [41 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Ossification Quality Score (Bony Ingrowth Assessed Via CT)
Description: The ossification quality score is an ordinal measure of quality of bone reabsorption that is divided into four progressive groups. Quality score 1 reflects "little or no bone ossification", Quality score 2 reflects "Some ossification; discontinuous or with a wide lucent rim", Quality score 3 reflects "Ossification with a thin lucent rim", and Quality score 4 reflects "Good ossification; border of tract vague". For this study, Quality scores 1 and 2 will be merged (defined as low quality ossification) as will Quality scores 3 and 4 (defined as high quality ossification).
  The proportion of suture anchors graded as having high quality ossification versus low quality ossification will be compared between the two groups to determine if there is a significant difference between Healicoil and Twinfix anchors in regards to quality of ossification.
Time Frame: 2 years
Population: The Ossification Quality Score will be assessed for each anchor implanted into a study subjects' shoulder. Because many subjects have more than one rotator cuff suture anchor implanted, the overall number of units analyzed will be greater than the overall number of participants analyzed.
Measure: Count of Units; unit: Suture Anchors
Units Other Than Participants: Suture Anchors
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
Number analyzed (Participants) | 26 | 26
Number analyzed (Suture Anchors) | 57 | 60
Suture Anchors
  Number of High Quality Ossification Anchors | 42 | 36
  Number of Low Quality Ossification Anchors | 15 | 24

2. Secondary Outcome: Number of Participants With a Rotator Cuff Re-tear
Description: Repair failure rate (Defined as number of subjects with a re-tear) determined by ultrasound 6 months after surgery.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
Number analyzed (Participants) | 26 | 26
Participants | 6 | 2

3. Secondary Outcome: Visual Analogue Pain Scale
Description: The Visual Analogue Pain Scale (VAS) measures the patient-reported level of pain at the two-year follow-up. The scale runs from 0 to 10, with "0" indicating no pain and "10" indicating extreme pain. The lower the VAS Pain level, the better the outcome in regards to level of pain.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
Number analyzed (Participants) | 26 | 26
score on a scale | 1.2 (1.3) | 1.8 (1.9)

4. Secondary Outcome: Function at Two Years as Measured by Western Ontario Rotator Cuff Index (WORC), PENN Shoulder Score (PENN), Single Assessment Numeric Evaluation (SANE), and EuroQol-5D (EQ-5D)
Description: Outcomes at Two Years on the following:
  * Western Ontario Rotator Cuff Index (WORC): developed to help understand the particular signs, symptoms, and functional limitations associated with rotator cuff tendinopathy. The outcome is measured on a scale of 0 to 100, with 100 being the best outcome and 0 being the worst.
  * PENN Shoulder Score (PENN): The PENN is a 100-point shoulder-specific self-report questionnaire evaluating pain, satisfaction, and shoulder function. The outcome is measured on a scale of 0 to 100, with 100 being the best outcome and 0 being the worst.
  * Single Assessment Numeric Evaluation (SANE): A single question that asks "How would you rate your shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?" 0 indicates an abnormal shoulder, whereas 100% indicates a perfectly normal shoulder.
  * Euroqol-5D (EQ-5D): The EQ-5D is a patient-reported overall health questionnaire, with 100 indicating "The best health you can imagine" and
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
Number analyzed (Participants) | 26 | 26
score on a scale
  SANE | 84.2 (20.9) | 86.7 (13.9)
  WORC | 78.7 (25.2) | 84.6 (13.5)
  PENN | 88.0 (13.6) | 88.6 (10.4)
  EQ-5D | 83.3 (16.3) | 87.3 (7.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected and assessed from time of surgery to two year final study follow-up
Arm/Group | HEALICOIL Regenesorb | Twinfix Ultra HA
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HEALICOIL Regenesorb (N=26) | Twinfix Ultra HA (N=26)
Loose biceps suture anchor (Surgical and medical procedures) | 0 (0) | 1 (1) — Loose anchored required revision surgery of the biceps.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT02350647/Prot_SAP_000.pdf